CLINICAL TRIAL: NCT05609149
Title: Risk Criteria Based on MRI Features Outperform Radiographic TNM Staging in Neoadjuvant Treatment Decisions for Patients With Rectal Cancer:A Single-Center, Open-Label, Retrospective, Observational Cohort Study
Brief Title: MRI Features in Neoadjuvant Treatment Decisions for Patients With Rectal Cancer
Status: Completed | Type: Observational
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yanhong Deng, Professor, Sun Yat-sen University
Other Study IDs: GIHSYSU-30
Record Dates: First submitted 2022-11-04; First posted 2022-11-08 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Rectal Cancer
Keywords: Rectal cancer; Neoadjuvant treatment; Mesorectal fascia; Extramural vascular invasion
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- T3 Rectal cancer: Patients with T3 rectal cancer who underwent curative surgery.
  Interventions: Procedure: total mesorectal excision

INTERVENTIONS:
Procedure: total mesorectal excision — patients must underwent total mesorectal excision

SUMMARY:
This study investigates whether risk criteria based on MRI features could identify a cohort of patients with a good prognosis among those recommended for preoperative treatment by NCCN guidelines to avoid preoperative treatment with the likely good survival outcomes by primary surgery and more accurately indicate the response to the treatment and predict prognosis after neoadjuvant treatmen than radiographic TNM staging in the patients who received neoadjuvant therapy.

DETAILED DESCRIPTION:
There is a lack of international consensus on the choice of preoperative treatment for patients with rectal cancer. Existing guidelines decide whether to administer preoperative therapy to patients with rectal cancer mainly based on the TNM system developed by AJCC/UICC, however, radiographic TNM staging is unsatisfactory in predicting the prognosis of patients with rectal cancer, due to inflammatory and fibrotic responses TNM re-staging is less accurate than pre-treatment. Studies have shown that high-resolution magnetic resonance imaging(MRI) accurately predicted pathologic findings such as CRM involvement, EMVI and TD and patients with MRI-detected CRM involvement, EMVI and TD are at risk for local and distant recurrence as well as poor overall survival. This retrospective study is designed to was to evaluate whether risk criteria based on MRI features can be used as a basis for neoadjuvant treatment decisions and more accurately indicate the response to the treatment and predict prognosis after neoadjuvant treatment than radiographic TNM staging. Patients with MRI-detected circumferential resection margin (CRM) involvement, extramural venous invasion (EMVI), or tumor deposits (TD) were defined as MRI high-risk.

ELIGIBILITY:
Inclusion Criteria:

1. Underwent primary rectal adenocarcinoma resection
2. Received MRI scan before surgery
3. Willing and able to provide written informed consent for participation in this study.
4. Treatment-naive patients with histological or cytological documentation of rectal adenocarcinoma (<12 cm from the anal verge).
5. Clinical stage of T3Nx or T1-3N+ at initial diagnosis
6. Non-complicated primary tumor (complete obstruction, perforation, bleeding).
7. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.

Exclusion Criteria:

1. Treated with transanal local excision
2. with distant metastases at the time of initial diagnosis
3. Subjects with a history of a prior malignancy within the past 5 years, except for adequately treated basal cell or squamous cell skin cancer.
4. Subjects with a history of any arterial thrombotic event within the past 6 months. This includes angina (stable or unstable), myocardial infarction (MI), Transient Ischemic Attacks (TIA), or cerebralvascular accident (CVA).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Rectal cancer patients with T3Nx or T1-3N+ at initial diagnosis.
Sampling Method: Non-Probability Sample
Enrollment: 480 (Actual)
Dates: Start 2016-10-30 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2022-11-02 (Actual)

PRIMARY OUTCOMES:
3-year event-free survival rate | 3 years after the surgery

SECONDARY OUTCOMES:
3-year overall survival rate | 3 years after the surgery
Local recurrence | 3 years after the surgery
  Defined as an intrapelvic recurrence following a primary rectal cancer resection, with or without distal metastasis.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of colorectal surgery, the Sixth Affiliated Hospital, Sun Yat-Sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided
Anonymous data may be provided upon reasonable request